CLINICAL TRIAL: NCT06213454
Title: Transversus Abdominis Plane Block Compared to Local Anesthetic Wound Infiltration in Gynecologic Oncology Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-1099; UW23039 (Other: UWCCC); NCI-2023-10464 (Registry Identifier: NCI CTRP); Protocol Version 7/17/2024 (Other: UW Madison); A532820 (Other: UW Madison)
Record Dates: First submitted 2024-01-09; First posted 2024-01-19 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Analgesia; Surgery
Keywords: laparotomy
MeSH Terms: conditions — Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: This is a randomized, unblinded, single-center trial testing the hypothesis that surgeon-initiated wound infiltration with local anesthetic is non-inferior in providing postoperative pain control when compared with preoperative TAP analgesia.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- TAP Block plus Laparotomy (Active Comparator)
  Interventions: Drug: TAP Anesthesia
- Laparotomy plus Local Wound Anesthetic (Active Comparator)
  Interventions: Drug: Surgeon-Initiated Local Anesthetic

INTERVENTIONS:
Drug: TAP Anesthesia — ultrasound guided TAP block, 133 mg of liposomal bupivacaine and 15 mL of 0.25% bupivacaine deposited into the TAP on each side for a total of two injections
  Other Names: bupivacaine; liposomal bupivacaine
  Arms: TAP Block plus Laparotomy
Drug: Surgeon-Initiated Local Anesthetic — 266 mg of liposomal bupivacaine and 30 mL of 0.25% bupivacaine diluted in 130 mL of normal saline (160 mL of solution), 40 mL fascial injection and 40 mL skin injection on either side of the wound
  Arms: Laparotomy plus Local Wound Anesthetic

SUMMARY:
This study is being done to see if preoperative transversus abdominis plane (TAP) analgesia will provide similar postoperative pain control, hospital length of stay, and postoperative outcomes compared to surgeon-initiated wound infiltration with local anesthetic in participants undergoing laparotomy for gynecologic indications.

DETAILED DESCRIPTION:
Primary Objective

* To evaluate the effects of preoperative TAP analgesia compared to surgeon-initiated wound infiltration with local anesthetic on pain control in subjects undergoing laparotomy.

Secondary Objectives

* To evaluate the effects of preoperative TAP analgesia compared to surgeon-initiated wound infiltration with local anesthetic on subject-rated perception of pain in subjects undergoing laparotomy.
* To evaluate the effects of preoperative TAP analgesia compared to surgeon-initiated wound infiltration with local anesthetic on length of hospital stay in subjects undergoing laparotomy.
* To evaluate the effects of preoperative TAP analgesia compared to surgeon-initiated wound infiltration with local anesthetic on postoperative anti-emetic use and number of recorded episodes of emesis in subjects undergoing laparotomy.
* To evaluate the effects of preoperative TAP analgesia compared to surgeon-initiated wound infiltration with local anesthetic on return of bowel function in subjects undergoing laparotomy.
* To evaluate the effects of preoperative TAP analgesia compared to surgeon-initiated wound infiltration with local anesthetic on subject satisfaction in subjects undergoing laparotomy.
* To evaluate the effects of preoperative TAP analgesia compared to surgeon-initiated wound infiltration with local anesthetic on postoperative complications in subjects undergoing laparotomy.
* To evaluate the effects of preoperative TAP analgesia compared to surgeon-initiated wound infiltration with local anesthetic on readmission rates in subjects undergoing laparotomy.
* To evaluate the cost of care associated with TAP analgesia compared to surgeon-initiated wound infiltration with local anesthetic on readmission rates in subjects undergoing laparotomy.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document
* Patients undergoing exploratory laparotomy via midline vertical skin incision for gynecologic indications at UW Hospital and Clinics
* Patients must be >18 years old
* English speaking (able to provide consent and complete questionnaires)
* Patients must have the ability to understand visual and verbal pain scales
* Patients must be eligible for TAP block placement. This will be confirmed during preoperative visit with the primary surgeon. Patient's are not eligible if they have allergies to the anesthetic medications or have had prior abdominal reconstructive surgery that would alter their abdominal wall anatomy in a way where the block would not be expected to be effective.

Exclusion Criteria:

* Known allergy to local anesthetics.
* Known history of chronic pain disorders and/or chronic opioid use defined as greater than 10mg of PO morphine or equivalent used daily for at least 30 days prior to enrollment.
* Patient has a history of opioid dependence requiring rehabilitation or the use of opioid antagonists.
* Patients with a planned exploration with biopsies (no organs removed) will be excluded from the study.
* Individuals who are pregnant, lactating or planning on becoming pregnant during the study.
* Significant liver disease that would inhibit prescription of opioids.
* Significant kidney disease that would inhibit administration of gabapentin.
* Not suitable for study participation due to other reasons at the discretion of the investigators.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Total opioid use measured in oral morphine equivalents for the first 24 hours post-surgery | 24 hours post-surgery
  Total opioid use measured in oral morphine equivalents for the first 24 hours post-surgery (including intraoperative and Post Anesthesia Care Unit (PACU) opioid utilization).

SECONDARY OUTCOMES:
Mean postoperative pain score for the first 24 hours post-surgery | 24 hours post-surgery
  Mean postoperative pain score for the first 24 hours post-surgery, measured by the Numeric Rating Scale (NRS), which rates pain on a 0-10 scale (collected routinely on the post-operative floor). Higher numbers indicate worse pain.
Length of hospital stay, measured in whole hours from admission to PACU to time of discharge order placement | estimated to be up to 3 days
Post-operative anti-emetic use | estimated to be up to 3 days
  A study team member will review the patient's medical chart to record the number of times an anti-emetic was given to the subject.
Number of recorded episodes of emesis | estimated to be up to 3 days
  A study team member will review the patient's medical chart to record number of times the hospital staff observed a participant vomit.
Return of bowel function measured in whole hours from completion of surgery to passage of flatus | estimated to be up to 3 days
Participant Satisfaction at Postoperative Visit measured by two pain questions from the QoR-15 Patient Reported Outcomes Survey Score | post-operative visit (up to 60 days)
  Scores are from 0-10 where 0 is pain all of the time and 10 is pain none of the time.
Readmission rate measured by readmission in the 30 days following surgery | up to 30 days
Cost of care measured by aggregate cost of hospitalization following discharge from surgical hospital stay | estimated to be up to 3 days
Summary of Post-operative Complications | up to 30 days post-operatively
  Postoperative complications, as defined by urinary tract infections, thromboembolic events, pneumonia, blood transfusion, cardiac events, falls, and electrolyte disturbances will be summarized by type and number of complications.
Time to First Ambulation measured in hours | estimated to be within 72 hours post-surgery
  A study team member will review the participant's medical chart to record the interval (in hours) from completion of surgery to first ambulation after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Sumer Wallace, MD, Principal Investigator — UW Carbone Cancer Center
Locations (1):
- University of Wisconsin Hospitals and Clinics (UWHC), Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No